CLINICAL TRIAL: NCT02586233
Title: A Phase 1b/2, Multi-Center, Double-Blind (Principal Investigators and Study Subjects Blinded, Sponsor Unblinded), Placebo-Controlled, Randomized, Single-Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of DS-1040b in Subjects With Acute Ischemic Stroke
Brief Title: Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of DS-1040b in Subjects With Acute Ischemic Stroke
Acronym: ASSENT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DS1040-A-U103; 2015-001824-43 (EudraCT Number)
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Results first posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-08

CONDITIONS: Acute Ischemic Stroke; Thrombotic Disease
Keywords: Acute Ischemic Stroke; Thrombotic disease; DS-1040b
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DS-1040b (Experimental): Participants who will be randomized to receive intravenous (IV) infusion of DS-1040b ranging from 0.6 mg to 9.6 mg.
  Interventions: Drug: DS-1040b
- Placebo (Placebo Comparator): Participants who will be randomized to receive intravenous (IV) infusion of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS-1040b — DS-1040b for IV infusion (0.6 mg to 9.6 mg) over 6-hour period
  Other Names: Experimental product
  Arms: DS-1040b
Drug: Placebo — 0.9% sodium chloride (placebo comparator) for IV infusion over 6-hour period
  Arms: Placebo

SUMMARY:
This is a Phase 1b/2, double-blind (study participants and Investigators), placebo-controlled, randomized, single-ascending dose, multi-center study to assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DS-1040b in participants with Acute Ischemic Stroke (AIS).

ELIGIBILITY:
Inclusion Criteria:

* Has a clinical diagnosis of acute ischemic stroke (including lacunar stroke/infarct) supported by computed topography or magnetic resonance imaging to rule out alternative cause for presenting symptoms
* Has onset of stroke symptoms within 4.5 to 12 hours before initiation of study drug administration - for subjects with a stroke upon waking, time of symptom onset is the last time the subject was known to be well
* Has a NIHSS score of ≥ 2 (for Cohorts 1-5) and ≥ 5 (for Cohort 6)
* Has Low dose heparin or low molecular weight heparin at a preventive dose are allowed from 24 hours after treatment start completion and after confirmation of no intracranial bleeding on the 24-hours repeat brain imaging.
* Is a Cohort 6 participant who is treated or anticipated to be treated with intra-arterial therapy (IAT) for ischemic stroke at the time of randomization (for enrollment in the IAT subgroup)
* Has given written informed consent to participate in the study prior to participating in any study-related procedures - depending on country-specific practice, written informed consent may be acceptable from legally authorized representative
* Has given a separate written informed consent for collecting a blood sample for genotyping

Exclusion Criteria:

* Is a Cohort 1-5 participant who has been treated or is going to be treated with tissue plasminogen activator (tPA) and/or endovascular thrombectomy during current stroke
* Is a Cohort 6 participant treated or anticipated to be treated with tPA during current stroke
* Has evidence of intracranial hemorrhage on non-contrast computed tomography (CT/CAT) scan or magnetic resonance imaging (MRI)
* Has symptoms of subarachnoid hemorrhage, even with normal imaging
* Has an Alberta Stroke Program Early CT Score (ASPECTS) <6
* Has prior non-traumatic intracranial hemorrhage (excluding microhemorrhages observed in imaging)
* Has known arteriovenous malformation or aneurysm
* Has evidence of active bleeding
* Has platelet count less than 100,000
* Has International Normalized Ratio greater than 1.7
* Has used unfractionated heparin within 24 hours prior to treatment and has an elevated partial thromboplastin time
* Has used a non-vitamin K antagonist oral anticoagulant such as dabigatran, rivaroxaban, apixaban, or other factor Xa inhibitors within 24 hours before treatment
* Has used fondaparinux or low molecular weight heparin at an anticoagulation dose within 24 hours prior to treatment
* Has anticipated use of an anticoagulation dose of heparin, or fondaparinux or low molecular weight heparin, or nonvitamin K antagonist oral anticoagulant such as dabigatran, rivaroxaban, apixaban, or other factor Xa inhibitors within 48 hours after completion of study drug treatment (low dose heparin or low molecular weight heparin at a preventive dose are allowed from 24 hours after treatment completion and after confirmation of no intracranial bleeding on the 24 hours repeat brain imaging. In Cohort 6, heparin treatment associated with IAT is allowed.)
* Has blood pressure > 185/110 mmHg, or requires aggressive medication to maintain blood pressure below this limit (routine medical treatment including IV drug treatment is allowed to lower the blood pressure below this limit)
* Has had intracranial surgery, clinically significant head trauma (in the opinion of Principal Investigator), Alteplase treatment, or a previous stroke within 1 month
* Has had major surgery within 14 days
* Has had gastrointestinal or genitourinary bleeding in the last 21 days
* Has had a lumbar puncture (or epidural steroid injection) within 14 days
* Has had a preexisting disability classified by modified Rankin Scale (mRS) > 2
* Has an estimated glomerular filtration rate < 60 mL/min/1.73 m^2
* Has baseline hemoglobin < 10.5 g/dL
* Has a positive pregnancy test
* Is currently participating in another investigational study or has participated in an investigational drug study within 30 days or 5 half-lives of that investigational drug prior to administration of the study drug
* Is an employee or an immediate family member of an employee of the Sponsor, the Contract Research Organization (CRO), or the Site
* Has any other condition the investigator determines would preclude participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (55):
- United States (16):
  - University of South Alabama USA Health System, Mobile, Alabama
  - UCLA Medical Center Stroke Network, Los Angeles, California
  - UC Health Memorial Hospital, Colorado Springs, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - JFK Neuroscience Institute, Edison, New Jersey
  - Icahn School Medicine at Mount Sinai, New York, New York
  - Duke University Health System, Durham, North Carolina
  - OSU - Wexner Medical Center, Columbus, Ohio
  - Oregon Health Sciences University Hospital, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Palmetto Health, USC School of Medicine, Columbia, South Carolina
  - Chattanooga Center for Neurologic Research, Chattanooga, Tennessee
  - Houston Methodist, Houston, Texas
- Australia (4):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital Neurology Dept., Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Czechia (2):
  - St. Annes University Hospital, Brno
  - Vitkovicka nemocnice a.s. Zaluzanskeho, Ostrava Vitkovice
- France (3):
  - CHRU Besançon - Hôpital Jean Minjoz, Besançon
  - Hôpital Pellegrin - CHU Bordeaux, Bordeaux
  - CHRU Lille - Hôpital Roger Salengro, Lille
- Germany (3):
  - Klinikum Altenburger Land, Altenburg
  - Universittsklinikum Essen AR Klinik fr Neurologie, Essen
  - Klinikum der Johann Wolfgang Goethe-Universitat, Frankfurt am Main
- Italy (6):
  - Ospedale di Citta di Castello, Città di Castello
  - Ospedale di Branca Largo Unita d'Italia, Gubbio
  - Ospedale Guglielmo da Saliceto Via Taverna, Piacenza
  - Ospedaliero di Albenga - Pietra Ligure Dept Neurology, Pietra Ligure
  - Azienda Ospedaliero Universitaria, Pisa
  - Ospedale Borgo Trento, Verona
- Slovakia (2):
  - Svet zdravia a.s.,Vseobecna nemocnica Rimavska Sobota, Rimavská Sobota
  - NsP Spisska Nova Ves, Spišská Nová Ves
- South Korea (3):
  - Pusan National University Hospital, Busan
  - Seoul National University Bundang Hospital, Seongnam-si
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital de la santa creu i sant pau C, Barcelona
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Clinico Universitario Lozano Blesa de Zaragoza, Zaragoza
- Taiwan (4):
  - Chang Gung Memorial Hospital-Linkou Branch, Taoyuan District, Hsien
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - University College Hospitals NHS Foundation Trust, London, England
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Salford Royal Hospital, Salford
  - Royal Stoke University Hospital, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 106 participants who met all inclusion criteria and no exclusion criteria were randomized to treatment at a total of 78 clinic sites (46 in Europe, 19 in the United States, 7 in Asia, 5 in Australia, and 1 in Canada). Of the 106 participants randomized, 101 participants received treatment.
Pre-assignment Details: The study consisted of 6, sequential, ascending-dose cohorts. Participants were randomized to either DS-1040b or placebo in a 3:1 ratio.
Groups:
- Cohort 1: DS-1040b 0.6 mg: Participants who received a single intravenous infusion of DS-1040b 0.6 mg.
- Cohort 2: DS-1040b 1.2 mg: Participants who received a single intravenous infusion of DS-1040b 1.2 mg.
- Cohort 3: DS-1040b 2.4 mg: Participants who received a single intravenous infusion of DS-1040b 2.4 mg.
- Cohort 4: DS-1040b 4.8 mg: Participants who received a single intravenous infusion of DS-1040b 4.8 mg.
- Cohort 5: DS-1040b 7.2 mg: Participants who received a single intravenous infusion of DS-1040b 7.2 mg.
- Cohort 6: DS-1040b 9.6 mg: Participants who received a single intravenous infusion of DS-1040b 9.6 mg.
- Placebo: Participants who received a single intravenous infusion of placebo.
Period: Overall Study
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg | Placebo
Started | 7 | 7 | 13 | 17 | 18 | 18 | 26
Completed | 7 | 5 | 13 | 17 | 16 | 16 | 24
Not Completed | 0 | 2 | 0 | 0 | 2 | 2 | 2
Not completed — Randomized but did not receive treatment | 0 | 1 | 0 | 0 | 0 | 2 | 2
Not completed — Death | 0 | 1 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographics and baseline characteristics were assessed in the Safety Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg | Placebo | Total
Number analyzed (Participants) | 7 | 6 | 13 | 17 | 18 | 16 | 24 | 101
Age, Categorical [Count of Participants; unit: Participants] — Population: Age data were missing for participants in some cohorts.
  Participants
    number analyzed (Participants) | 6 | 6 | 12 | 15 | 17 | 16 | 23 | 95
    <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 2 | 3 | 8 | 8 | 9 | 9 | 13 | 52
    >=65 years | 4 | 3 | 4 | 7 | 8 | 7 | 10 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age data were missing for participants in some cohorts.
  years
    number analyzed (Participants) | 6 | 6 | 12 | 15 | 17 | 16 | 23 | 95
    (all) | 68.2 (7.8) | 68.2 (10.2) | 62.7 (9.7) | 69.1 (11.1) | 65.8 (11.7) | 64.8 (12.8) | 62.2 (12.3) | 65.2 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5 | 6 | 8 | 6 | 11 | 41
  Male | 4 | 4 | 8 | 11 | 10 | 10 | 13 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 4 | 8 | 2 | 3 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 2 | 0 | 1 | 4 | 10
  White | 6 | 4 | 11 | 11 | 10 | 13 | 17 | 72
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Summary of Treatment-Emergent Adverse Event Reported by >10% of Participants Following Ascending Doses of DS-1040b and a Placebo in Participants With Acute Ischemic Stroke
Description: Treatment-emergent adverse event (TEAE) is defined as an adverse event that emerges during the treatment period (from first dose date until 30 days after the last dosing date), having been absent at predose; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pre-dose state, when the adverse event is continuous.
Time Frame: Baseline up to 90 days post last dose, up to 3 years 11 months
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- All DS-1040b: All participants who received a single intravenous infusion of DS-1040b.
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg | All DS-1040b | Placebo
Number analyzed (Participants) | 7 | 6 | 13 | 17 | 18 | 16 | 77 | 24
Participants
  Any TEAE | 5 | 5 | 10 | 15 | 14 | 14 | 63 | 18
  Hypokalaemia | 1 | 2 | 2 | 0 | 2 | 2 | 9 | 6
  Constipation | 1 | 2 | 3 | 1 | 5 | 2 | 14 | 5
  Insomnia | 0 | 0 | 1 | 0 | 1 | 3 | 5 | 5
  Hypertension | 0 | 0 | 1 | 3 | 1 | 0 | 5 | 3
  Anxiety | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 3
  Hyperglycaemia | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3
  Dyslipidaemia | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3
  Thrombocytopenia | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Vomiting | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Pyrexia | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
  Vitamin B12 deficiency | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Headache | 3 | 1 | 2 | 2 | 1 | 4 | 13 | 2

2. Secondary Outcome: Summary of Pharmacokinetic (PK) Parameter Maximum (Peak) Observed Plasma Concentration (Cmax) of DS-1040b Following Ascending Doses in Participants With Acute Ischemic Stroke
Description: The PK parameter of Maximum (Peak) Observed Plasma Concentration (Cmax) of DS-1040b was calculated from the plasma concentrations of DS-1040b using non-compartmental analysis
Time Frame: Predose, 0.5, 3, 6, 9, 12, 24, 48, 72, and 96 hours postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg
Number analyzed (Participants) | 5 | 6 | 13 | 16 | 17 | 10
ng/mL | 10.09 (3.26) | 26.95 (9.39) | 61.28 (35.67) | 729.76 (1661.06) | 191.06 (59.60) | 203.70 (41.49)

3. Secondary Outcome: Summary of Pharmacokinetic Parameter Area Under the Concentration Versus Time Curve From Zero to Last Quantifiable Concentration Sampling Point (AUClast) of DS-1040b Following Ascending Doses in Participants With Acute Ischemic Stroke
Description: The PK parameter of Area Under the Concentration Versus Time Curve from Zero to Last Quantifiable Concentration Sampling Point of DS-1040b was calculated from the plasma concentrations of DS-1040b using non-compartmental analysis
Time Frame: Predose, 0.5, 3, 6, 9, 12, 24, 48, 72, and 96 hours postdose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg
Number analyzed (Participants) | 5 | 6 | 13 | 16 | 17 | 10
ng*h/mL | 69.74 (16.19) | 219.83 (95.16) | 447.75 (199.97) | 2611.87 (4471.65) | 1489.21 (460.78) | 1700.24 (346.43)

4. Secondary Outcome: Summary of Pharmacokinetic Parameter Terminal Half-life (t1/2) of DS-1040b Following Ascending Doses in Participants With Acute Ischemic Stroke
Description: The PK parameter of Terminal Half-life of DS-1040b was calculated from the plasma concentrations of DS-1040b using non-compartmental analysis in patients with available sample for the analysis.
Time Frame: Pre-dose, 0.5, 3, 6, 9, 12, 24, 48, 72, and 96 hours post-dose
Population: Pharmacokinetic parameters were assessed in the Pharmacokinetic Analysis Set, except for terminal half-life which was assessed in patients with available sample for the analysis.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg
Number analyzed (Participants) | 4 | 2 | 7 | 8 | 14 | 8
h | 2.59 (0.46) | 4.14 (0.17) | 10.50 (15.02) | 36.68 (25.94) | 33.37 (14.71) | 35.86 (10.98)

5. Secondary Outcome: Summary of Activated Form of Thrombin-activatable Fibrinolysis Inhibitor (TAFIa) Following Ascending Doses of DS-1040b and a Placebo in Participants With Acute Ischemic Stroke
Description: The enzymatic activity of thrombin-activatable fibrinolysis inhibitor was assessed using the Stago Coagulation Analyzer.
Time Frame: Baseline and 6 hours postdose
Population: TAFIa activity was assessed in the Pharmacodynamic Analysis Set.
Measure: Mean (Standard Deviation); unit: mean percentage of TAFIa activity
Groups:
- Cohort 6: DS-1040b 9.6 mg (Non-IAT): Participants who received a single intravenous infusion of DS-1040b 9.6 mg (non-intra-arterial thrombectomy).
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg (Non-IAT) | Placebo
Number analyzed (Participants) | 7 | 6 | 13 | 17 | 18 | 10 | 24
mean percentage of TAFIa activity
  Baseline: number analyzed (Participants) | 7 | 5 | 13 | 16 | 17 | 9 | 19
  Baseline | 96.7 (23.7) | 97.8 (17.5) | 100.4 (21.6) | 105.1 (23.4) | 108.1 (30.5) | 112.6 (27.2) | 100.9 (20.8)
  6 h postdose: number analyzed (Participants) | 6 | 6 | 10 | 16 | 17 | 9 | 21
  6 h postdose | 93.5 (26.6) | 98.8 (27.2) | 86.7 (16.7) | 75.9 (20.9) | 72.9 (22.6) | 73.9 (14.4) | 104.1 (24.7)

6. Secondary Outcome: Summary of Changes From Baseline at Day 30 in National Institute of Health Stroke Scale (NIHSS) Score Following Ascending Doses of DS-1040b and a Placebo in Participants With Acute Ischemic Stroke
Description: The National Institute of Health Stroke Scale (NIHSS) quantifies stroke severity based on weighted evaluation findings. The score for each ability is a number between 0 and 4, with 0 being normal functioning and 4 being completely impaired. The patient's NIHSS score is calculated by adding the number for each element of the scale; 42 is the highest score possible. In the NIHSS, the higher the score indicates more impairment (worse outcome) in a stroke patient.
Time Frame: 30 days post dose
Population: NIHSS stroke scale scores were assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg | All DS-1040b | Placebo
Number analyzed (Participants) | 7 | 6 | 13 | 17 | 18 | 16 | 77 | 24
units on a scale | -3.7 (2.21) | -3.0 (2.00) | -3.5 (1.71) | -2.06 (1.06) | -3.4 (2.70) | -6.2 (3.08) | -3.9 (2.56) | -3.6 (4.27)

7. Secondary Outcome: Percentage of Participants With a Modified Rankin Scale (mRS) Score of 0 to 2 Following Ascending Doses of DS-1040b and a Placebo in Participants With Acute Ischemic Stroke
Description: The modified Rankin scale (mRS) is a commonly used disability scale derived from the Rankin scale that is used to measure the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The level of disability following a stroke is assessed via a scale from 0 to 6, where 0 is no symptoms at all and 6 indicates death. Higher scores indicate worse outcome. The percentage of participants with an mRS score of 0 to 2 at Day 5 (baseline) and Day 90 is being reported.
Time Frame: Day 5 (baseline) and Day 90 post dose
Population: Modified Rankin scale scores were assessed in the Safety Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg | All DS-1040b | Placebo
Number analyzed (Participants) | 7 | 6 | 13 | 17 | 18 | 16 | 77 | 24
percentage of participants
  Day 5: number analyzed (Participants) | 6 | 5 | 13 | 17 | 18 | 15 | 74 | 24
  Day 5 | 66.7 | 40.0 | 76.9 | 82.4 | 72.2 | 53.3 | 68.9 | 54.2
  Day 90: number analyzed (Participants) | 7 | 5 | 13 | 17 | 16 | 16 | 74 | 24
  Day 90 | 85.7 | 60.0 | 76.9 | 82.4 | 93.8 | 68.8 | 79.7 | 75.0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from baseline up to 30 days post last dose, up to 3 years 11 months.
Description: A TEAE is defined as an adverse event that: emerges during the treatment period (from first dose date until 30 days after the last dosing date), having been absent at predose; or reemerges during treatment, having been present at baseline but stopped prior to treatment; or worsens in severity after starting treatment relative to the pre-dose state, when the adverse event is continuous.
Arm/Group | Cohort 1: DS-1040b 0.6 mg | Cohort 2: DS-1040b 1.2 mg | Cohort 3: DS-1040b 2.4 mg | Cohort 4: DS-1040b 4.8 mg | Cohort 5: DS-1040b 7.2 mg | Cohort 6: DS-1040b 9.6 mg | All DS-1040b | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/6 | 0/13 | 0/17 | 2/18 | 0/16 | 3/77 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/6 | 0/13 | 1/17 | 2/18 | 2/16 | 10/77 | 4/24
Other Adverse Events (participants affected / at risk) | 5/7 | 5/6 | 10/13 | 15/17 | 14/18 | 14/16 | 63/77 | 18/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DS-1040b 0.6 mg (N=7) | Cohort 2: DS-1040b 1.2 mg (N=6) | Cohort 3: DS-1040b 2.4 mg (N=13) | Cohort 4: DS-1040b 4.8 mg (N=17) | Cohort 5: DS-1040b 7.2 mg (N=18) | Cohort 6: DS-1040b 9.6 mg (N=16) | All DS-1040b (N=77) | Placebo (N=24)
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Spinal cord infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DS-1040b 0.6 mg (N=7) | Cohort 2: DS-1040b 1.2 mg (N=6) | Cohort 3: DS-1040b 2.4 mg (N=13) | Cohort 4: DS-1040b 4.8 mg (N=17) | Cohort 5: DS-1040b 7.2 mg (N=18) | Cohort 6: DS-1040b 9.6 mg (N=16) | All DS-1040b (N=77) | Placebo (N=24)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 4 | 2
Hyperfibrinogenaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 6 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 5 | 2 | 14 | 5
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 6 | 2
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 4 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Influenza-like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Infusion-site phlebitis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1 | 4 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyuria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 3 | 1 | 6 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 1 | 4 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Post-procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Biopsy bone (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 4 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Fluid imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 0 | 2 | 2 | 9 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Circadian rhythm sleep disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasticity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Neurological decompensation (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Neurological symptom (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paraesthesia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 2 | 1 | 4 | 13 | 2
Stroke in evolution (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 3 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 5 | 5
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Urethral pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 3 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 3 | 1 | 0 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02586233/Prot_SAP_000.pdf